CLINICAL TRIAL: NCT05027399
Title: Nursing Teleconsultation for Patients With Heart Failure Due to Hypersensitive, Chagasic or Idiopathic
Brief Title: Nursing Teleconsultation for Patients With Heart Failure
Acronym: NurTHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Monitoring by teleconsultation
Record Dates: First submitted 2021-07-28; First posted 2021-08-30 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Nurse; Teleconsultation; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: After filtering this patient database, following the inclusion and exclusion criteria, will be performed randomization in two groups of 30 participants, randomization will be stratified by two variables, Age and Ejection Fraction, using the Jamovi statistical software. Group A will be composed of the participants who will have intervention, that is, the patients will receive fortnightly follow-up in nursing telephone consultation concurrently with follow-up usual outpatient clinic and group B (control) will be composed of the participants who will have no intervention and will continue to monitor according to the institution's routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Consultations will be carried out via video call, every 15 days for a period of 3 months, with a total of 6 telephone consultations that will have in order to clarify doubts about the CI, the monitoring of possible clinical signs of instability and help in adapting or creating strategies for better adherence to therapy.
  Interventions: Behavioral: Nursing teleconsultation for lifestyle changes
- Control Group (No Intervention): Will be composed by the participants who will have no intervention and will continue to monitor according to the institution's routine.

INTERVENTIONS:
Behavioral: Nursing teleconsultation for lifestyle changes — Guidance on better medication adherence, monitoring of signs and symptoms of exacerbation of heart failure, guidance on the need for fluid restriction.
  Arms: Intervention Group

SUMMARY:
The incidence and prevalence of heart failure are increasing and represent a large portion of hospitalizations in Brazil, are also associated with high rates of morbidity, mortality and costs for the service of health. Such data, added to the current scenario of the pandemic caused by COVID-19, reveal the need for changes in clinical practice, so that health care is more effective and cost-effective and reaches patients without exposing them to risks. Thus, the application of nursing interventions through of telephone technology, which has strong evidence of effectiveness found in the literature, has become an alternative for the implementation of clinical interventions. Objective: Evaluate the effectiveness of nursing consultations performed remotely in improving quality of life and adherence to therapy of patients with HF due to cardiomyopathy of different etiologies. Method: The study will have as methodological framework the randomized clinical trial, with the recruitment of 60 volunteers with a diagnosis of chagasic HF, Hypertensive or Idiopathic, who are monitored at the outpatient clinic of Clinical Unit of Cardiomyopathies and Aortic Diseases or Clinical Unit of Hypertension, InCor-HCFMUSP, included by drawing lots into two groups. group A (n=30) will be monitored in biweekly nursing consultations by a period of three months added to the outpatient follow-up, and group B (n = 30) will follow the usual outpatient follow-up. Hypothesis: Patients HF carriers who periodically make telephone consultations of nursing have better quality of life and better therapeutic adherence when compared to patients who only have regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients already registered in a database of the Clinical Unit of Cardiomyopathies and Aortic Diseases, InCor - HCFMUSP and Clinical Hypertension Unit - HCFMUSP, in outpatient follow-up for more than a year;
* Stroke Volume < 40% and >25%

Exclusion Criteria:

* Patientes with Pacemaker, Defibrillators, Implantable and Cardiac Resynchronization Therapy
* Listed in heart transplant queue
* Not having technological devices that allow the teleconsultation to be carried out
* Psychic inability to understand the questionnaires and answer the questions asked by the interviewer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
Improvement in the quality of life of patients who receive teleconsultations with a nurse | 3 months
  To analyze this result, the questionnaire Minnesota Living with Heart Failure Questionnaire (MLHFQ) validated in portuguese language will be used. Zero is the minimum value and 105 maximum value, The lower score, represents a better patient's quality of life.
Improvement in the therapeutic adhesion of patients who receive teleconsultations with a nurse | 3 months
  To analyze this result, the questionnaire European Heart Failure Self-Care Behaviour Scale (EHFScBS) validated in portuguese language will be used. 12 is the minimum value and 60 maximum value, The lower score, represents a better self care.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor), Hospital das Clinicas do HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No share plan

REFERENCES:
- [Background] Gomes BR, Bocchi EA. Quality of Life in Heart Failure: An Important Goal in Treatment. Arq Bras Cardiol. 2020 Jan;114(1):33-34. doi: 10.36660/abc.20190741. No abstract available. PMID 32049167
- [Background] Fang JC, Ewald GA, Allen LA, Butler J, Westlake Canary CA, Colvin-Adams M, Dickinson MG, Levy P, Stough WG, Sweitzer NK, Teerlink JR, Whellan DJ, Albert NM, Krishnamani R, Rich MW, Walsh MN, Bonnell MR, Carson PE, Chan MC, Dries DL, Hernandez AF, Hershberger RE, Katz SD, Moore S, Rodgers JE, Rogers JG, Vest AR, Givertz MM; Heart Failure Society of America Guidelines Committee. Advanced (stage D) heart failure: a statement from the Heart Failure Society of America Guidelines Committee. J Card Fail. 2015 Jun;21(6):519-34. doi: 10.1016/j.cardfail.2015.04.013. Epub 2015 May 4. PMID 25953697
- [Background] Rutledge CM, Kott K, Schweickert PA, Poston R, Fowler C, Haney TS. Telehealth and eHealth in nurse practitioner training: current perspectives. Adv Med Educ Pract. 2017 Jun 26;8:399-409. doi: 10.2147/AMEP.S116071. eCollection 2017. PMID 28721113